CLINICAL TRIAL: NCT00894517
Title: A Study Evaluating the Effect of Botulinum Toxin Type A on Semen Quality in Patients With Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-091
Record Dates: First submitted 2009-05-05; First posted 2009-05-07 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-07

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin Type A (Experimental): OnabotulinumtoxinA (botulinum toxin Type A) 200U injected into the prostate on Day 1.
  Interventions: Biological: Botulinum Toxin Type A
- Placebo (saline) (Placebo Comparator): Placebo (saline) injected into the prostate on Day 1.
  Interventions: Drug: Placebo (saline)

INTERVENTIONS:
Biological: Botulinum Toxin Type A — OnabotulinumtoxinA (botulinum toxin Type A) 200U injected into the prostate on Day 1.
  Other Names: BOTOX®
  Arms: Botulinum Toxin Type A
Drug: Placebo (saline) — Saline injected into the prostate on Day 1.
  Arms: Placebo (saline)

SUMMARY:
This is a 24 week study evaluating the effects of botulinum toxin Type A on semen quality in patients with signs and symptoms of Benign Prostatic Hyperplasia (BPH).

ELIGIBILITY:
Inclusion Criteria:

* Symptoms due to an enlarged prostate
* Able to provide semen samples at required visits.

Exclusion Criteria:

* Previous use of any botulinum toxin for the treatment of any urological condition
* History of vasectomy
* History of undescended testicles or testicular trauma
* Subject who has not ejaculated for greater than 1 year
* History of prostate infection or any sexually transmitted disease, such as gonorrhea, within the previous 12 months
* History of bladder stones
* History of cancer in the prostate, testicles, or bladder
* Previous use of chemotherapy for cancer treatment
* History of urinary incontinence
* Previous prostate surgery

Ages: 45 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo (Normal Saline): Placebo (Normal saline) injected into the prostate on Day 1.
Period: Overall Study
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Started | 30 | 31
Completed | 28 | 26
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline) | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Customized [Number; unit: Participants]
  45 to 60 years | 20 | 25 | 45
  > 60 years | 10 | 6 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 31 | 61

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Total Sperm Count Per Ejaculate
Description: Sperm count per ejaculate was calculated based on the average of two semen samples collected 2 to 5 days apart at Baseline and at Week 12. Ejaculatory volume and sperm concentration were used to determine the total sperm count per ejaculate. A positive percent change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: Safety population included all randomized participants who received treatment.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Number analyzed (Participants) | 29 | 30
Percent change | 3.62 (56.773) | -12.22 (57.564)

2. Secondary Outcome: Change From Baseline in Log Transformed Sperm Concentration
Description: Sperm concentration was calculated based on the average of two semen samples collected 2 to 5 days apart at Baseline and at Week 12. Collected sperm samples were assessed using a CELL-VU® count chamber. The total number of sperm per 100 boxes on the chamber grid were counted. Sperm Concentration = total number of sperm counted in 100 boxes × dilution factor / 1 × 10^6 and is reported in millions per milliliter. Log transformation of the sperm concentration was used for analysis . The log transformed sperm concentration data has no units. A negative change from Baseline indicated a lower sperm concentration (worsening).
Time Frame: Baseline, Week 12
Population: Safety population included all randomized participants who received treatment.
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Number analyzed (Participants) | 29 | 30
Unitless
  Baseline | 3.77 (0.765) | 3.82 (0.814)
  Change from Baseline at Week 12 (n=29, 27) | -0.13 (0.599) | -0.23 (0.457)

3. Secondary Outcome: Change From Baseline in Ejaculatory Volume
Description: Ejaculatory volume was calculated using the average of two semen samples collected 2 to 5 days apart at Baseline and at Week 12. Ejaculatory volume was measured using a standard pipette (measuring device). A negative change from Baseline indicated worsening.
Time Frame: Baseline, Week 12
Population: Safety population included all randomized participants who received treatment.
Measure: Mean (Standard Deviation); unit: milliliters (mL)
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Number analyzed (Participants) | 29 | 30
milliliters (mL)
  Baseline | 2.30 (1.170) | 2.35 (1.267)
  Change from Baseline at Week 12 (n=29, 28) | -0.12 (0.813) | -0.09 (0.690)

4. Secondary Outcome: Change From Baseline in Total Sperm Motility
Description: Sperm motility was calculated using the average of two semen samples collected 2 to 5 days apart at Baseline and at Week 12. Sperm motility was assessed using the CELL-VU chamber and was scored according to the World Health Organization criteria for sperm progression and motility. A total of at least 200 motile and immotile sperm were counted. A percent was determined by the calculation of motile sperm/total sperm count. A negative change from Baseline indicated a worsening.
Time Frame: Baseline, Week 12
Population: Safety population included all randomized participants who received treatment.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Number analyzed (Participants) | 29 | 30
Percent
  Baseline | 53.67 (14.214) | 55.15 (11.519)
  Change from Baseline at Week 12 (n=29, 28) | -1.50 (13.142) | -3.93 (14.167)

5. Secondary Outcome: Change From Baseline in Normal Sperm Morphology
Description: Sperm Morphology was evaluated using the average of two semen samples collected 2 to 5 days apart at Baseline and at Week 12. Normal sperm morphology was assessed from slide smears sent to a central reading facility. A positive change from Baseline indicated improvement.
Time Frame: Baseline, Week 12
Population: Safety population included all randomized participants who received treatment.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Number analyzed (Participants) | 29 | 30
Percent
  Baseline | 12.37 (3.503) | 14.14 (2.989)
  Change from Baseline at Week 12 (n=29, 28) | 0.36 (0.852) | 0.05 (1.240)

ADVERSE EVENTS:
Description: The safety population (all randomized and treated participants) was used to calculate the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | Botulinum Toxin Type A | Placebo (Normal Saline)
Serious Adverse Events (participants affected / at risk) | 0/29 | 3/30
Other Adverse Events (participants affected / at risk) | 18/29 | 12/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=29) | Placebo (Normal Saline) (N=30)
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Botulinum Toxin Type A (N=29) | Placebo (Normal Saline) (N=30)
Urinary tract infection (Infections and infestations) | 4 | 1
Haematuria (Renal and urinary disorders) | 2 | 2
Nephrolithiasis (Renal and urinary disorders) | 2 | 2
Dysuria (Renal and urinary disorders) | 2 | 0
Micturition urgency (Renal and urinary disorders) | 2 | 0
Haematospermia (Reproductive system and breast disorders) | 4 | 7
Ejaculation delayed (Reproductive system and breast disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.